CLINICAL TRIAL: NCT00275418
Title: Double-Blind Randomized Prospective Trial of Treatment With Natural Beta Carotene Vs. Placebo for Patients With Crohn's Disease in Remission
Brief Title: Beta Carotene From Natural Source for Patients With Non-Active Crohn's Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Beta Carotene 01
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 2006-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; remission; beta carotene
MeSH Terms: conditions — Crohn Disease

INTERVENTIONS:
Drug: beta carotene from Dunaliella algae

SUMMARY:
Many inflammatory disorders in the body are linked to oxidative tissue damage. Anti-oxidants that are present in many natural food sources may provide protection from such damage.

Beta carotene is an anti-oxidant vitamin present in many fruits and vegetables. The algae Dunaliella is particularly rich in beta carotene.

In this prospective trial we want to investigate whether beta carotene from Dunaliella may prevent exacerbations of Crohn's disease.

DETAILED DESCRIPTION:
Patients with documented Crohn's disease who are at least 2 months in remission (CDAI<150) will be randomized to receive 60 mg beta carotene/day vs. placebo for 1 year.

The study medication will be taken in addition to regular treatment for Crohn's disease.

The protocol includes 5 visits (months 0, 3, 6, 9, 12). Each visit lasts 30-60 minutes and includes a brief interview, standard questionnaires, physical examination, and blood tests.

Exacerbation of Crohn's disease is defined as CDAI>150. The study hypothesis is that less patients treated with beta carotene will suffer an exacerbation than patients treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients with documented Crohn's disease in remission (CDAI<150) for at least two months, age 17-75 years

Exclusion Criteria:

* active Crohn's disease (CDAI>150), partial bowel obstruction, impending surgery, pregnancy, serious other diseases

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2002-07

PRIMARY OUTCOMES:
CDAI score measured 3-monthly during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Lavy, MD, Principal Investigator — Technion, Haifa, Israel
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel